CLINICAL TRIAL: NCT03480152
Title: A Phase I/II Trial to Evaluate the Safety and Immunogenicity of a Messenger RNA (mRNA)-Based, Personalized Cancer Vaccine Against Neoantigens Expressed by the Autologous Cancer
Brief Title: Messenger RNA (mRNA)-Based, Personalized Cancer Vaccine Against Neoantigens Expressed by the Autologous Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Rosenberg, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 180074; 18-C-0074
Record Dates: First submitted 2018-03-27; First posted 2018-03-29 (Actual); Results first posted 2020-04-24 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Melanoma; Colon Cancer; Gastrointestinal Cancer; Genitourinary Cancer; Hepatocellular Cancer
Keywords: Metastatic Cancer; Immunotherapy; Tumor Regression; Cancer Vaccine; Gene Therapy
MeSH Terms: conditions — Melanoma; Colonic Neoplasms; Gastrointestinal Neoplasms; Urogenital Neoplasms; Liver Neoplasms; Neoplasm Metastasis | interventions — National Cancer Institute (U.S.)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/Phase - Escalating doses of mRNA vaccine (Experimental): Escalating doses of messenger ribonucleic acid (mRNA) vaccine
  Interventions: Biological: National Cancer Institute (NCI)-4650, a messenger ribonucleic acid (mRNA)-based, Personalized Cancer Vaccine
- 2/Phase II -MTD of mRNA vaccine established in Phase I (Experimental): Maximum tolerated dose (MTD) of messenger ribonucleic acid (mRNA) vaccine established in Phase I
  Interventions: Biological: National Cancer Institute (NCI)-4650, a messenger ribonucleic acid (mRNA)-based, Personalized Cancer Vaccine

INTERVENTIONS:
Biological: National Cancer Institute (NCI)-4650, a messenger ribonucleic acid (mRNA)-based, Personalized Cancer Vaccine — Patients will receive a messenger ribonucleic acid (mRNA)-based vaccine intramuscularly at two-week intervals for four cycles (one course of treatment). Patients may be vaccinated with a second and final course of treatment using the same vaccine dose. The second course may start approximately four weeks (plus or minus 2 weeks) from the last vaccine dose of the first course.

SUMMARY:
Background:

Exome sequencing can identify certain gene mutations in a person's tumor. This can then be used to create cancer treatments. In this study, researchers will make a treatment called a messenger ribonucleic acid (mRNA) vaccine. The vaccine might cause certain tumors to shrink.

Objective:

To see if the mRNA vaccine is safe and can cause metastatic melanoma or epithelial tumors to shrink.

Eligibility:

People 18-70 years old with metastatic melanoma or epithelial cancer

Design:

Participants will be screened under protocol 99-C-0128.

Participants will provide samples under protocol 03-C-0277:

Participants will provide a piece of their tumor from a previous surgery or biopsy.

Participants will have leukapheresis: Blood is removed through a needle in one arm and circulated through a machine that takes out the white blood cells. The blood is then returned through a needle in the other arm.

Participants will have many tests:

Scans and x-rays

Heart and lung function tests

Blood and urine tests

Participants will receive the mRNA vaccine every 2 weeks for up to 8 weeks. They will get the vaccine as an injection into the upper arm or thigh. They may receive a second course of vaccines if the study doctor determines it is needed.

Participants will have follow-up visits approximately 2 weeks after their final vaccine, then 1 month later, then every 1-2 months for the first year, and then once a year for up to 5 years. Each visit may take up to 2 days and include:

Physical exam

Blood tests

Scans

Leukapheresis at the first visit

DETAILED DESCRIPTION:
Background:

* Therapeutic vaccination against cancer has proven very challenging with little clinical benefit.
* Vaccines against non-viral tumors have mainly targeted differentiation antigens, cancer testis antigens, and overexpressed antigens. However, negative selection in the thymus against these normal non-mutated antigens severely limits the ability to generate high avidity anti-cancer T-cells. Such depletion can impair their antitumor activity and limit tumor elimination.
* The National Cancer Institute Surgery Branch (NCI-SB) has developed a pipeline for the identification of immunogenic T-cell epitopes derived from neoantigens.
* In recent studies, we identified the neoantigens recognized by tumor-infiltrating lymphocytes (TIL) that mediated regression in patients with metastatic melanoma. Using whole exome sequencing of a resected metastatic nodule followed by high throughput immunologic screening, we were able to demonstrate that tumor regressions were associated with the recognition by the administered TIL of unique somatic mutations that occurred in the cancer.
* We also found that TIL from 29 of 32 patients with a wide variety of metastatic gastrointestinal cancers contained lymphocytes that recognized unique mutations presented in that patient's cancer.
* We, therefore, aim to use this pipeline to identify immunogenic neoantigens and to predict for neoantigens binding the patient human leukocyte antigen (HLA) molecules from melanoma or epithelial cancer patients and to use these epitopes for a personalized therapeutic messenger ribonucleic acid (mRNA) vaccine.

Objectives

Primary objectives:

* Determine the clinical response rate in patients with metastatic melanoma, gastrointestinal or genitourinary cancers who receive NCI-4650
* Determine the safety of NCI-4650 in patients with metastatic melanoma, gastrointestinal or genitourinary cancers

Eligibility

* Age greater than or equal to 18 years and less than or equal to 70 years
* Evaluable metastatic melanoma, gastrointestinal, or genitourinary cancers refractory to standard of care treatment
* Metastatic cancer lesions suitable for surgical resection to perform whole exome sequencing and preparation of TIL

Design:

* Patients with metastatic cancer will undergo surgical resection of tumor followed by exome and RNA sequencing to identify expressed mutations. This will be conducted under the NCI-SB cell harvest protocol 03-C-0277. (Cell Harvest and Preparation for Surgery Branch Adoptive Cell Therapy Protocols).
* Immunogenic neoantigens will be identified from TIL by high throughput immunologic screening using long peptides and tandem minigenes covering all mutated epitopes.
* Up to 15 predicted neoantigens will be selected based on exome and RNA sequencing and their binding affinity to the patient HLA molecules.
* The mRNA vaccine will be manufactured and supplied as Current Good Manufacturing Practice (cGMP) product by ModernaTX, Inc.
* The patient will be vaccinated with mRNA containing epitopes from immunogenic neoantigens, predicted neoantigens and mutations in tumor suppressor or driver genes.
* The mRNA vaccine will be administered intramuscularly (IM) for four cycles every two weeks. A patient may receive a second course for a total of eight cycles given.
* Blood samples will be taken every two weeks (during the vaccination period) and at each follow-up visit, and patients will be monitored for the quantity and quality of circulating neoantigen-specific T-cells.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Measurable (per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria), metastatic melanoma, gastrointestinal, or genitourinary cancer with at least one lesion that is resectable. Only patients with metastatic gastrointestinal cancer will be eligible for enrollment on the Phase I portion of the study. Patients with metastatic melanoma, gastrointestinal, or genitourinary cancer will be eligible for enrollment on the Phase II portion of the study.
* Confirmation of diagnosis of metastatic cancer by the National Cancer Institute (NCI) Laboratory of Pathology.
* Patients with 3 or fewer brain metastases that are less than 1 cm in diameter and asymptomatic are eligible. Lesions that have been treated with stereotactic radiosurgery must be clinically stable for one month after treatment for the patient to be eligible. Patients with surgically resected brain metastases are eligible.
* Prior therapy with at least one first-line standard of care treatment or second-line treatment of proven effectiveness. Patients must have progressive disease after prior treatment. Prior first-or second-line treatments would include the following:

  * Patients with metastatic melanoma: Receipt of a checkpoint inhibitor as first-line therapy
  * Patients with metastatic melanoma with an activating mutation of KIT: Receipt of Imatinib
  * Patients with a BRAF V600 activating mutation: Receipt of appropriate targeted therapy
  * Patients with metastatic gastrointestinal cancer: Receipt of up to two forms of approved first- and/or second-line chemotherapy regimens
  * Patients with metastatic genitourinary cancers: Receipt of a first- or second-line therapy appropriate for their histologic subtype
* Age greater than or equal to 18 years and less than or equal to 70 years.
* Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 or 1.
* Serology

  * Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive may have decreased immune-competence and thus may be less responsive to the experimental treatment and more susceptible to its toxicities.)
  * Seronegative for hepatitis B antigen, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then the patient must be tested for the presence of antigen by reverse transcription polymerase chain reaction (RT-PCR) and be hepatitis C virus (HCV) ribonucleic acid (RNA) negative.
* Hematology

  * Absolute neutrophil count (ANC) > 1000/mm(3) without the support of growth factors.
  * White blood cell (WBC) greater than or equal to 3000/mm(3)
  * Platelet count greater than or equal to 100.000/mm(3)
  * Hemoglobin > 8.0 g/dl. Subjects may be transfused to reach this cut-off.
* Chemistry

  * Serum Alanine aminotransferase (ALT)/Aspartate aminotransferase (AST) less than or equal to 5.0 times upper limit of normal (ULN)
  * Serum creatinine <1.5 times ULN or measured creatinine clearance (calculated using Cockcroft-Gault formula) > 40 ml/min
  * Total bilirubin less than or equal to 2.0 mg/dl, except in patients with Gilbert's Syndrome, who must have a total bilirubin < 3.0 mg/dl.
* More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the immunization regimen, and patients' toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo).
* Ability of subject to understand and the willingness to sign a written informed consent document.
* Subjects must be co-enrolled on protocol 03-C-0277.

EXCLUSION CRITERIA:

* Pregnant or breastfeeding women who do not consent to stop breast-feeding while on study treatment and for 30 days after the use of the investigational vaccine where pregnancy is confirmed by a positive, rising human chorionic gonadotropin (hCG) laboratory test.

  * Women of child-bearing potential, defined as all women capable of becoming pregnant, unless they agree to use an appropriate method of contraception during dosing and for 120 days after the last dose (i.e., final vaccine). Effective contraception methods include a combination of any two of the following (unless method is abstinence or sterilization, in which only one method is required):

    * Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%). In case of use of oral contraception, women should have been stable on the same pill for a minimum of 6 months before taking study treatment.
    * Placement of an intrauterine device or intrauterine system.
    * Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.
    * Total abstinence
    * Female sterilization at least eight weeks before taking study treatment.
    * Male sterilization (at least six months prior to screening).
* Sexually active males must use a condom during intercourse during dosing and for 120 days after the last dose (i.e., final vaccine), and should not father a child in this period.
* Any systemic steroid therapy or other form of immunosuppressive therapy within 7 days of the first dose of the vaccine. A physiologic dose of systemic corticosteroids may be approved. Inhaled or topical steroids, and less than or equal to 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
* Active systemic infections requiring anti-infective treatment, coagulation disorders, or any other active or uncompensated major medical illnesses of the cardiovascular, respiratory, or immune system.
* Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
* Concurrent opportunistic infections (the experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
* Any vaccinations four weeks prior to the first vaccination cycle or live vaccines at any time during the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-05-18 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2019-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Rosenberg, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klein L, Hinterberger M, Wirnsberger G, Kyewski B. Antigen presentation in the thymus for positive selection and central tolerance induction. Nat Rev Immunol. 2009 Dec;9(12):833-44. doi: 10.1038/nri2669. PMID 19935803
- [Background] Bos R, Marquardt KL, Cheung J, Sherman LA. Functional differences between low- and high-affinity CD8(+) T cells in the tumor environment. Oncoimmunology. 2012 Nov 1;1(8):1239-1247. doi: 10.4161/onci.21285. PMID 23243587
- [Background] Abramson J, Giraud M, Benoist C, Mathis D. Aire's partners in the molecular control of immunological tolerance. Cell. 2010 Jan 8;140(1):123-35. doi: 10.1016/j.cell.2009.12.030. PMID 20085707
- [Derived] Cafri G, Gartner JJ, Zaks T, Hopson K, Levin N, Paria BC, Parkhurst MR, Yossef R, Lowery FJ, Jafferji MS, Prickett TD, Goff SL, McGowan CT, Seitter S, Shindorf ML, Parikh A, Chatani PD, Robbins PF, Rosenberg SA. mRNA vaccine-induced neoantigen-specific T cell immunity in patients with gastrointestinal cancer. J Clin Invest. 2020 Nov 2;130(11):5976-5988. doi: 10.1172/JCI134915. PMID 33016924

RESULTS

PARTICIPANT FLOW:
Recruitment Details: No participants were enrolled on Dose Level 1 - 0.04mg vaccine, nor Cohort 2a/2b, Arm 2, Phase II Maximum Tolerated Dose Arm/Group. Participants vaccination started on Dose Level 2 - 0.13 mg.
Pre-assignment Details: Two step registration process. Step One: Patient signed consent to create vaccine. Step Two: Once vaccine is available, patient screened for eligibility criteria. If eligibility criteria were met, registration and enrollment was completed and the patient was treated. One patient died between Step one and Step two and was not treated.
Groups:
- Cohort 1, Arm 1, Phase I - Dose Level 2 - 0.13mg: Gastrointestinal cancer patients receive 0.13mg of messenger ribonucleic acid (mRNA) vaccine as intramuscular (IM) injections on Days 0, 14, 28, and 42.
- Cohort 1, Arm 1, Phase I - Dose Level 3 - 0.39mg: Gastrointestinal cancer patients receive 0.39mg of messenger ribonucleic acid (mRNA) vaccine as intramuscular (IM) injections on Days 0, 14, 28, and 42.
- Cohort 2a/2b, Arm 2, Phase II Maximum Tolerated Dose: (2a) Melanoma and (2b) Gastrointestinal or Genitourinary cancer patients receive the maximum tolerated dose (MTD) of messenger ribonucleic acid (mRNA) vaccine established in Phase I.
Period: Phase I
Arm/Group | Cohort 1, Arm 1, Phase I - Dose Level 2 - 0.13mg | Cohort 1, Arm 1, Phase I - Dose Level 3 - 0.39mg | Cohort 2a/2b, Arm 2, Phase II Maximum Tolerated Dose
Started | 3 | 2 | 0
Received Intervention | 2 | 2 | 0
Completed | 2 | 2 | 0
Not Completed | 1 | 0 | 0
Not completed — Signed consent. Died before treatment. | 1 | 0 | 0
Period: Phase II
Arm/Group | Cohort 1, Arm 1, Phase I - Dose Level 2 - 0.13mg | Cohort 1, Arm 1, Phase I - Dose Level 3 - 0.39mg | Cohort 2a/2b, Arm 2, Phase II Maximum Tolerated Dose
Started | 0 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No baseline data was collected for the participant that signed consent for vaccine but died before treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1, Arm 1, Phase I - Dose Level 2 - 0.13mg | Cohort 1, Arm 1, Phase I - Dose Level 3 - 0.39mg | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (4) | 51 (6) | 46.5 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had a Clinical Response (Complete Response + Partial Response) to Treatment (Objective Tumor Regression)
Description: Clinical response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Complete Response (CR) is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. Partial Response (PR) is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. Stable Disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of diameters while on study. Progressive Disease (PD) is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
Time Frame: up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Arm 1, Phase I - Dose Level 2 - 0.13mg | Cohort 1, Arm 1, Phase I - Dose Level 3 - 0.39mg
Number analyzed (Participants) | 2 | 2
Participants
  Complete Response | 0 | 0
  Partial Response | 0 | 0
  Stable Disease | 0 | 0
  Progressive Disease | 2 | 2
  Not Evaluable | 0 | 0

2. Primary Outcome: Number of Non-Serious Adverse Events Probably Related to Treatment
Description: Here is the number of non-serious adverse events probably related to treatment assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0).
Time Frame: During treatment and up to 30 days after the first follow- up evaluation (at the second follow-up evaluation)
Measure: Number; unit: adverse events
Groups:
- Cohort 1, Arm 1, Phase I - Dose Level 2 - 0.13mg Starting Dose: Gastrointestinal Cancer patients receive 0.13mg of messenger ribonucleic acid (mRNA) vaccine as intramuscular (IM) injections on Days 0, 14, 28, and 42.
Arm/Group | Cohort 1, Arm 1, Phase I - Dose Level 2 - 0.13mg Starting Dose | Cohort 1, Arm 1, Phase I - Dose Level 3 - 0.39mg
Number analyzed (Participants) | 2 | 2
adverse events
  Nausea | 0 | 2
  Vomiting | 0 | 1

3. Secondary Outcome: Number of Participants With an Increase in the Quantity and Quality of Circulating Antigen-specific T Cells
Description: Participants blood samples were assessed by fluorescence-activated cell sorting (FACS), enzyme-linked immune absorbent (ELISA)-spot and human soluble cluster of differentiation 137 (CD137) (4-1BB) upregulation assays. Differences of 2-3 fold in these assays over the baseline measures are indicative of true biologic difference.
Time Frame: Approximately 2 weeks after last vaccine
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Arm 1, Phase I - Dose Level 2 - 0.13mg | Cohort 1, Arm 1, Phase I - Dose Level 3 - 0.39mg
Number analyzed (Participants) | 2 | 2
Participants | 2 | 2

4. Other Pre Specified Outcome: Number of Participants With Non-Serious Adverse Events Regardless of Attribution
Description: Here is the count of participants with non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence.
Time Frame: Date treatment consent signed to date off study, approximately 11 months and 4 days.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1, Arm 1, Phase I - Dose Level 3 - 0.39mg: Gastrointestinal cancer patients receive 0.39mg of messenger ribonucleic acid (mRNA) vaccine as intramuscular injections (IM) on Days 0, 14, 28, and 42.
Arm/Group | Cohort 1, Arm 1, Phase I - Dose Level 2 - 0.13mg | Cohort 1, Arm 1, Phase I - Dose Level 3 - 0.39mg
Number analyzed (Participants) | 2 | 2
Participants | 2 | 2

5. Other Pre Specified Outcome: Number of Dose Limiting Toxicities (DLT)
Description: A DLT is all Grade 3 or greater toxicities related to the messenger ribonucleic acid vaccine with exception of Grade 3 fever, Grade 3 pruritic/itching, Grade 3 fatigue, Grade 3 metabolic laboratory abnormalities without significant clinical sequela that resolves to Grade 2 or less within 7 days, Grade 3 autoimmune toxicity that resolves to Grade 2 or less in 7 days and events that are clearly related to the patient's disease.
Time Frame: Up to 21 days after the first vaccination
Measure: Number; unit: toxicities
Arm/Group | Cohort 1, Arm 1, Phase I - Dose Level 2 - 0.13mg | Cohort 1, Arm 1, Phase I - Dose Level 3 - 0.39mg
Number analyzed (Participants) | 2 | 2
toxicities | 0 | 0

6. Other Pre Specified Outcome: Maximum Tolerated Dose (MTD
Description: A MTD is the highest dose at which ≤1 of 6 patient's experienced a dose limiting toxicity (i.e., All Grade 3 or greater toxicities related to the messenger ribonucleic acid vaccine with exception of Grade 3 fever, Grade 3 pruritic/itching, Grade 3 fatigue, Grade 3 metabolic laboratory abnormalities without significant clinical sequela that resolves to Grade 2 or less within 7 days, Grade 3 autoimmune toxicity that resolves to Grade 2 or less in 7 days and events that are clearly related to the patient's disease.) or the highest dose level studied if DLT's are not observed at any of the dose levels.
Time Frame: Up to 21 days after the first vaccination
Population: MTD was not reached.
Arm/Group | Cohort 1, Arm 1, Phase I - Dose Level 2 - 0.13mg
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 11 months and 4 days.
Description: Two step registration process. Step One: Patient signed consent to create vaccine. Step Two: Once vaccine is available, patient screened for eligibility criteria. If eligibility criteria were met, registration and enrollment was completed and the patient was treated. One patient died between Step one and Step two and was not treated.
Arm/Group | Cohort 1, Arm 1, Phase I - Dose Level 2 - 0.13mg | Cohort 1, Arm 1, Phase I - Dose Level 3 - 0.39mg
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1, Arm 1, Phase I - Dose Level 2 - 0.13mg (N=2) | Cohort 1, Arm 1, Phase I - Dose Level 3 - 0.39mg (N=2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2) — Possibly related to research.
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) — Possibly related to research.
Fatigue (General disorders) | 1 (2) | 2 (5)
Fever (General disorders) | 0 (0) | 2 (2)
Flu like symptoms (General disorders) | 1 (2) | 1 (1)
Injection site reaction (General disorders) | 2 (8) | 2 (4)
Pain (General disorders) | 1 (1) | 0 (0)
Shingles (Infections and infestations) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, excoriation to the head of penis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Chills (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-23): https://cdn.clinicaltrials.gov/large-docs/52/NCT03480152/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-28): https://cdn.clinicaltrials.gov/large-docs/52/NCT03480152/ICF_001.pdf